CLINICAL TRIAL: NCT01267903
Title: A Phase Ia Clinical Trial for Inactivated Vaccine(Vero Cell) Against EV71 in Chinese Healthy Young Adults and Children
Brief Title: A Clinical Trial for Inactivated Vaccine(Vero Cell) Against EV71 in Chinese Healthy Young Adults and Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Collaborators: Bejing Vigoo Biological Co., LTD (Industry)
Responsible Party: Zhu Fengcai, Jiangsu Provincial Center for Diseases Control and Prevention
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JSVCT003
Record Dates: First submitted 2010-12-28; First posted 2010-12-29 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-01

CONDITIONS: Hand, Foot and Mouth Disease
Keywords: Vaccines Adverse Reaction
MeSH Terms: conditions — Hand, Foot and Mouth Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 320U /0.5ml in young adults (Experimental): inactivated vaccine(vero cell) against EV71 of 320U /0.5ml in 20 young adults aged 16-22 years old on day0,28
  Interventions: Biological: vaccine against EV71 of 320U/0.5ml
- 640U /0.5ml in young adults (Experimental): inactivated vaccine(vero cell) against EV71 of 640U /0.5ml in 20 young adults aged 16-22 years old on day0,28
  Interventions: Biological: vaccine against EV71 of 640U/0.5ml
- 160U /0.5ml in children (Experimental): inactivated vaccine(vero cell) against EV71 of 160U /0.5ml in 20 children aged 5-15 years old on day0,28
  Interventions: Biological: vaccine against EV71 of 160U/0.5ml
- 320U /0.5ml in children (Experimental): inactivated vaccine(vero cell) against EV71 of 320U /0.5ml in 20 children aged 6-15 years old on day0,28
  Interventions: Biological: vaccine against EV71 of 320U/0.5ml
- 640U /0.5ml in children (Experimental): inactivated vaccine(vero cell) against EV71 of 640U /0.5ml in 20 children aged 6-15 years old on day0,28
  Interventions: Biological: vaccine against EV71 of 640U/0.5ml

INTERVENTIONS:
Biological: vaccine against EV71 of 320U/0.5ml — inactivated vaccine(vero cell) against EV71 of 320U/0.5ml on day0,28,modern medicines
  Arms: 320U /0.5ml in young adults
Biological: vaccine against EV71 of 640U/0.5ml — inactivated vaccine(vero cell) against EV71 of 640U/0.5ml on day0,28
  Arms: 640U /0.5ml in young adults
Biological: vaccine against EV71 of 160U/0.5ml — inactivated vaccine(vero cell) against EV71 of 160U/0.5ml on 0,28 day
  Arms: 160U /0.5ml in children
Biological: vaccine against EV71 of 320U/0.5ml — inactivated vaccine(vero cell) against EV71 of 320U/0.5ml on day0,28
  Arms: 320U /0.5ml in children
Biological: vaccine against EV71 of 640U/0.5ml — inactivated vaccine(vero cell) against EV71 of 640U/0.5ml on day0,28
  Arms: 640U /0.5ml in children

SUMMARY:
Hand, foot, and mouth disease (HFMD) is a common viral illness in infants and children caused by viruses that belong to the enterovirus genus of the picornavirus family. Although most HFMD cases do not result in serious complications, outbreaks of HFMD caused by enterovirus 71 (EV71) can present with a high rate of neurological complications, including meningoencephalitis, pulmonary complications, and can even cause infant death. HFMD caused by EV71 has become a major emerging infectious disease in Asia and the highly pathogenic potential of EV71 clearly requires the attention of world medical community.

The development of vaccine against EV71 is active and ongoing in Asian countries now. Several studies have examined the effectiveness of inactivated viral vaccines against EV71 in animal model. A wide range of experimental EV71 vaccine approaches have been studied including heat-inactivated or formaldehyde-inactivated virion, EV71 virus-like particles (VLP) , VP1 recombinant protein ,VP1 DNA vaccine , VP1 peptide-based vaccine targeting the neutralizing domain, bacterial or viral vector expressing VP1, and a Vero cell-adapted live attenuated virus. Furthermore, neutralizing antibodies against EV71 have been suggested as one of the most important factors in prevention of the severe EV71 infection. Recently, an inactivated vaccine(vero cell) against EV71 has been licensed by SFDA in China, this clinical trial phase Ia is armed to evaluate safety and tolerance in Chinese healthy adults and children.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged from 5 to 22 years old as established by medical history and clinical examination
* The subjects or their guardians are able to understand and sign the informed consent
* Had never received the vaccine against EV71
* Subjects who can and will comply with the requirements of the protocol

Exclusion Criteria:

* Subject that has a medical history of HFMD
* subject that has a medical history of any of the following: allergic history, or allergic to any ingredient of vaccine
* Family history of seizures or progressive neurological disease
* Family history of congenital or hereditary immunodeficiency
* Women of pregnancy, lactation or about to be pregnant in 60 days
* Autoimmune disease or immunodeficiency
* Bleeding disorder diagnosed by a doctor or significant bruising or bleeding difficulties with IM injections or blood draws
* Any prior administration of administration of immunoglobulins

Ages: 5 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2011-01; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
to evaluate the safety of EV71 vaccine in Chinese healthy adults and children | 28 days after the first vaccination
  to evaluate the Adverse reactions of EV71 vaccine in Chinese healthy adults and children
to evaluate the safety of EV71 vaccine in Chinese healthy adults and children | 28 days after the second vaccination
  to evaluate the Adverse reactions of EV71 vaccine in Chinese healthy adults and children

SECONDARY OUTCOMES:
to evaluate the seroconversion rate of Antinuclear antibodies in serum after first vaccination | 28 days after the first vaccination
  to evaluate the seroconversion rate of Antinuclear antibodies in serum 28 days after first vaccination
to evaluate the seroconversion rate of Antinuclear antibodies in serum after second vaccination | 28 days after second vaccination
  to evaluate the seroconversion rate of Antinuclear antibodies in serum 28 days after second vaccination
to evaluate the abnormity change of live and kidney function indexes in serum after first vaccination | 3 days after first vaccination
  to evaluate the abnormity change of live and kidney function indexes in serum 3 days after first vaccination
to evaluate the abnormity change of live and kidney function indexes in serum after second vaccination | 3 days after second vaccination
  to evaluate the abnormity change of live and kidney function indexes in serum 3 days after second vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Fengcai Zhu, Master, Principal Investigator — Jiangsu Provincial Center for Diseases Control and Prevention

REFERENCES:
- [Derived] Meng FY, Li JX, Li XL, Chu K, Zhang YT, Ji H, Li L, Liang ZL, Zhu FC. Tolerability and immunogenicity of an inactivated enterovirus 71 vaccine in Chinese healthy adults and children: an open label, phase 1 clinical trial. Hum Vaccin Immunother. 2012 May;8(5):668-74. doi: 10.4161/hv.19521. Epub 2012 May 1. PMID 22634437